## Oral human administration of red grape polyphenol in nickel-mediated allergic contact dermatitis: an in vitro study

Statistical analysis was performed using GraphPad Prism 5.02 (GraphPad Software, USA). Differences were considered statistically significant for p<0.05.

In order to compare statistical differences between two groups data obtained were analyzed by two-way ANOVA followed by a Bonferroni post hoc test. Differences within groups were determined by a paired Student *t* test